CLINICAL TRIAL: NCT07289542
Title: A Randomized, Blinded and Placebo-Control Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of Lyophilized Respiratory Syncytial Virus mRNA Vaccine in Adults Aged 50 Years or Above
Brief Title: Phase II Clinical Trial of Lyophilized Respiratory Syncytial Virus mRNA Vaccine in Adults Aged 50 Years or Above
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Collaborators: Abogen Biosciences (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABO1105-201
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Dose level A in adults aged 50 years or above (Experimental): Single injection of Dose level A of ABO1105
  Interventions: Biological: ABO1105
- Group 2: Dose level B in adults aged 50 years or above (Experimental): Single injection of Dose level B of ABO1105
  Interventions: Biological: ABO1105
- Group 3: Placebo control in adults aged 50 years or above (Placebo Comparator): Single injection of placebo on Day 0
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ABO1105 — Formulation for injection
  Arms: Group 1: Dose level A in adults aged 50 years or above; Group 2: Dose level B in adults aged 50 years or above
Drug: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Group 3: Placebo control in adults aged 50 years or above

SUMMARY:
The primary objective of this study is to evaluate the immunogenicity and safety of a single injection of two dose levels of ABO1105 in adults aged 50 years or above.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the Informed Consent Form (ICF) approved by the Ethics Committee and agree to participate in the trial before undergoing any trial procedures.
2. Healthy adults ≥50 years of age, participants with underlying diseases that are stably controlled may be accepted.
3. Willing to and physically able to communicate with the investigators, understand and comply with protocol required follow-up, simple self-observation and recording using the Diary Card.
4. Male participants (and their female partners) and female participants of childbearing potential agree to continue effective contraception through 3 months following vaccination.

Exclusion Criteria:

1. Presence of one or more respiratory symptoms within 7 days prior to vaccination, lasting for at least 24 hours.
2. Acute illness or fever within 3 days prior to vaccination, or use of anti-inflammatory, anti-allergy, antibiotic, or antiviral medications due to physical discomfort.
3. Laboratory-confirmed history of RSV infection within the past 12 months, or previous vaccination with a respiratory syncytial virus vaccine.
4. Clinically significant abnormal vital signs, including but not limited to:

   * Resting pulse rate <50 beats per minute or >100 beats per minute, participants with resting pulse between 100 to 110 without significant symptoms, such as palpitations, chest tightness, dizziness and fatigue, will be accepted.
   * Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg for participants aged 50-59, or systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg for participants aged ≥60
   * Body mass index (BMI) ≥30 kg/m²
5. Female participants known to be pregnant or breastfeeding, or positive pregnancy test for women of childbearing potential.
6. History of allergy to any ingredients of the investigational products, or severe allergic reactions to other vaccines, foods, or medications.
7. Use or planned use of any vaccine other than the investigational products through 30 days prior to and 30 days after vaccination in this trial.
8. Current participation in another clinical trial within 30 days prior to vaccination or planned participation before the end of this trial.
9. Clinician-diagnosed coagulation abnormalities.
10. Known medical history or diagnosis confirming the subject has a condition affecting immune system function.
11. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or presence of any condition that may increase the risk of myocarditis or pericarditis.
12. Severe or uncontrolled respiratory, cardiovascular, neurological, hematological, lymphatic, hepatic, renal, metabolic, or skeletal diseases; known severe congenital malformations; developmental disorders; or clinically diagnosed severe chronic conditions that may affect trial outcomes.
13. Current infectious period of any communicable disease, acute infection, or acute phase of chronic infection, or ongoing anti-tuberculosis treatment; or prior positive test for hepatitis B surface antigen, hepatitis C virus antibody, or Treponema pallidum antibody.
14. Past or current diagnosis of neurological or psychiatric disorders, or family history of neurological/psychiatric disorders; or other neurological conditions deemed unsuitable for trial participation by the investigator.
15. Long-term use of immunosuppressants or immunomodulators within 6 months prior to vaccination, excluding topical medications. Topical medications should not exceed recommended doses or induce systemic exposure.
16. Treatment with immunoglobulins and/or blood products or blood donation through 3 months prior to and 3 months after vaccination in this trial.
17. Suspected or known alcohol dependence or drug abuse, which may affect safety assessment or trial compliance.
18. Planned long-term or permanent relocation away from the trial site area before trial completion.
19. Investigators, sponsors, and contract research organization (CRO) staff directly involved in the trial.
20. Other circumstances deemed unsuitable for trial participation by the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum RSV Neutralizing Antibodies (Abs) | Up to Day 30
Geometric Mean Increase versus Postbaseline/Baseline Ab Titers | Up to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Baise Center For Disease Control & Prevention, Baise City, Baise, China

IPD SHARING:
Plan to Share IPD: No